CLINICAL TRIAL: NCT05983354
Title: Oral v. Parenteral Medications for the Emergency Management of Acute Migraine: a Pilot Randomized Control Trial
Brief Title: Oral Medications for the Management of Acute Migraine Headache in the Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Sciences North Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-016
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: Acute Migraine Headache
Keywords: emergency department; migraine; metoclopramide
MeSH Terms: conditions — Emergencies; Migraine Disorders | interventions — Metoclopramide; Ibuprofen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment will be randomly assigned using a random number generator by an independent research assistant who is not involved in data collection. Contents of treatment will be known only to the research pharmacist and this information will be stored remotely from the ED; patients, administering nurses and treating physicians will be blind to the treatment group, as well the research assistants collecting outcome data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral medications (Experimental): 10 mg oral metoclopramide, 400 mg oral ibuprofen with 2 x 50 ml NS administered over 15 minutes.
  Interventions: Drug: Oral metoclopramide and ibuprofen
- IV medications (Active Comparator): 2 x placebo tablets, 10 mg metoclopramide in 50 cc NS and 10 mg ketorolac in 50 ml NS administered over 15 min.
  Interventions: Drug: Intravenous metoclopramide and ketorolac

INTERVENTIONS:
Drug: Oral metoclopramide and ibuprofen — 10 mg oral metoclopramide, 400 mg oral ibuprofen with 2 x 50 ml normal saline IV administered over 15 minutes.
  Other Names: Maxeran, Reglan
  Arms: Oral medications
Drug: Intravenous metoclopramide and ketorolac — 10 mg of metoclopramide IV in 50 ml normal saline, 10 mg ketorolac IV in 50 ml normal saline administered over 15 minutes, with 2 placebo tablets.
  Other Names: Maxeran, Reglan, Toradol
  Arms: IV medications

SUMMARY:
The goal of this pilot randomized control trial is to assess the feasibility of our patient recruitment and data collection strategy ahead of a full scale RCT investigating the efficacy of oral v. parenteral medications in the management of acute migraine headaches in the emergency department. Patients will be randomly assigned to receive either (A) standard medical therapy for the treatment of acute migraine headache (metoclopramide and ketorolac IV) and oral placebo or (B) oral metoclopramide and ibuprofen with normal saline IV. Primary outcome measures are recruitment rate and improvement in pain score at 60 minutes from medication administration.

DETAILED DESCRIPTION:
Objectives

The planned study is a pilot study designed to assess the feasibility of our recruitment and data collection strategy. The primary feasibility outcome will be recruitment rate, which is defined as the proportion of eligible patients approached who are successfully recruited over the proposed 6-month pilot study period. Our secondary feasibility outcomes are (a) proportion of eligible patients approached and (b) rate of attrition during the study period.

Our preliminary primary outcome will be improvement in pain from baseline to 60 minutes after medication administration using the visual analogue scale (Bijur et al. 2008). Preliminary secondary outcomes will include headache relief and freedom from headache at 2 h, the need for rescue medication, ED length of stay and return to ED within 24h of discharge. The frequency of adverse effects, including gastrointestinal upset, patient-reported restlessness or dystonic reaction and fatigue, will be assessed.

Design

In this parallel, noninferiority, double-blind randomised control pilot study, eligible patients presenting to the emergency department with a chief complaint of headache will be randomly assigned with an allocation ratio of 1:1 to receive one of 2 treatments: intravenous ketorolac (10 mg) and metoclopramide (10 mg) v. oral ibuprofen (400 mg) and metoclopramide (10 mg). Dosing was selected to reflect the lowest effective doses recommended for emergency department management of migraine headaches (Friedman et al. 2011, Motov et al. 2017). The study will last 6 months at which time it will stop.

Study population

Patients between the ages of 18 and 64 presenting to the ED with a chief complaint of headache will be eligible to participate in the study. Exclusion criteria include vomiting or inability to tolerate oral medications at the time of medication administration, focal neurologic symptoms, head trauma within 14 days, history of renal disease, contraindication to NSAIDs including pregnancy or concurrent use of blood thinners, hypersensitivity reaction to any of the study medications, or >15 headache days per month.

Study procedures

Treatment will be assigned using a random number generator. Contents of treatment, which will be identical in appearance, will be known only to the research pharmacist and this information will be stored remotely from the ED. Administering nurses and treating physicians will be blind to the treatment group, as will patients and research assistants collecting outcome data.

Data collection

Data will be collected using patient interviews immediately prior to medication administration and repeated at 1 and 2 hours after medication administration. A chart review will then be conducted to check for return visits within 24 h of ED discharge.

Enrolment:

Based on sample size calculations, 55 patients will be enrolled.

Statistical procedures:

Primary and secondary feasibility outcomes will be reported as the proportion of patients approached who were recruited, proportion of eligible patients approached and the proportion who withdrew consent during the study period +/- 95% CI.

ELIGIBILITY:
Inclusion Criteria:

- Presentation to emergency department with headache

Exclusion Criteria:

* Vomiting or unable to tolerate PO at tie of med admin
* Focal neurologic symptoms
* Head trauma within 14d
* Pregnancy
* Concurrent use of blood thinners
* Hypersensitivity reaction to any of the study medications
* >14 HA days per month

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Proportion of eligible patients presenting to ED who are successfully recruited
Pain relief | 60 minutes
  Change in visual analogue scale (0-10 where 0 is no pain and 10 is maximal pain) from baseline to 60 minutes after medication administration

SECONDARY OUTCOMES:
Proportion of eligible patients approached | 6 months
  Proportion of all eligible patients who were approached by research assistants
Rate of attrition during the study period | 24 hours
  Number of patients recruited to study who ended participation during study period
Pain relief at 2 hours | 120 minutes
  Change in visual analogue scale from baseline to 120 minutes after medication administration
Freedom from headache | 60 minutes
  Patients who report complete resolution of headache at 60 minutes from medication administration
Need for rescue medication | 24 h
  Additional medications administered by treating physician after 60 minutes
Emergency department length of stay | 24 hours
  Time from initial physician assessment to discharge
Return to emergency department | 24 hours
  Patients who were registered again to the ED within 24 hours of discharge
Adverse reactions | 24 hours
  Any adverse reaction reported during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ohle, MBBCh, Principal Investigator — Health Sciences North Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azzopardi TD, Brooks NA. Oral metoclopramide as an adjunct to analgesics for the outpatient treatment of acute migraine. Ann Pharmacother. 2008 Mar;42(3):397-402. doi: 10.1345/aph.1K481. Epub 2008 Feb 19. PMID 18285561
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Burch RC, Loder S, Loder E, Smitherman TA. The prevalence and burden of migraine and severe headache in the United States: updated statistics from government health surveillance studies. Headache. 2015 Jan;55(1):21-34. doi: 10.1111/head.12482. Erratum In: Headache. 2015 Feb;55(2):356. PMID 25600719
- [Background] Burch R, Rizzoli P, Loder E. The prevalence and impact of migraine and severe headache in the United States: Updated age, sex, and socioeconomic-specific estimates from government health surveys. Headache. 2021 Jan;61(1):60-68. doi: 10.1111/head.14024. Epub 2020 Dec 21. PMID 33349955
- [Background] Friedman BW, Mulvey L, Esses D, Solorzano C, Paternoster J, Lipton RB, Gallagher EJ. Metoclopramide for acute migraine: a dose-finding randomized clinical trial. Ann Emerg Med. 2011 May;57(5):475-82.e1. doi: 10.1016/j.annemergmed.2010.11.023. Epub 2011 Jan 12. PMID 21227540
- [Background] Motov S, Yasavolian M, Likourezos A, Pushkar I, Hossain R, Drapkin J, Cohen V, Filk N, Smith A, Huang F, Rockoff B, Homel P, Fromm C. Comparison of Intravenous Ketorolac at Three Single-Dose Regimens for Treating Acute Pain in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2017 Aug;70(2):177-184. doi: 10.1016/j.annemergmed.2016.10.014. Epub 2016 Dec 16. PMID 27993418
- [Background] Yeh WZ, Blizzard L, Taylor BV. What is the actual prevalence of migraine? Brain Behav. 2018 Jun;8(6):e00950. doi: 10.1002/brb3.950. Epub 2018 May 2. PMID 30106228